CLINICAL TRIAL: NCT02058758
Title: Quantitative Methods for Supplementing Contrast-Enhanced Magnetic Resonance Imaging of Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1312M4621; R21CA179070 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-02-10 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Magnetic resonance spectroscopy; Diffusion weighted imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Device: Magnetic Resonance Imaging
  Interventions: Device: Magnetic Resonance Imaging
- Breast Cancer Patients: Device: Magnetic Resonance Imaging
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — MRI scanning with novel acquisition, reconstruction, and/or analysis methods.

SUMMARY:
Contrast-enhanced magnetic resonance imaging (CE-MRI) is now established as the most accurate non-invasive imaging modality for characterizing breast cancer. CE-MRI has a very high sensitivity because the intravenous MR contrast agent highlights regions with increased vascularization and vascular permeability compared to normal breast tissues and benign lesions.

DETAILED DESCRIPTION:
Contrast-enhanced magnetic resonance imaging (CE-MRI) is now established as the most accurate non-invasive imaging modality for characterizing breast cancer. CE-MRI has a very high sensitivity because the intravenous MR contrast agent highlights regions with increased vascularization and vascular permeability compared to normal breast tissues and benign lesions. While research continues on improving the specificity of CE-MRI, several other MR techniques that do not require an exogenous contrast agent have been shown to provide valuable information that can improve the characterization of breast cancers. These techniques include magnetic resonance spectroscopy (MRS), diffusion-weighted imaging, and water T2 relaxometry. The long-term goal of this study is to develop these techniques to produce quantitative MR-based biomarkers that can be used to supplement or possibly supplant the information provided by CE-MRI. This project seeks to facilitate the advancement of these advanced, non-contrast techniques. This study uses a piggyback design, in which subjects who are already scheduled to receive a CE-MRI study are invited to receive an additional 10-20 minutes of scanning to help develop these novel methods. This efficient design allows for the refinement and assessment of these new techniques with a minimum of risk and inconvenience to the patient. With these proposed improvements, these techniques may lead to quantitative biomarkers that can guide critical clinical questions in treatment response, diagnosis, staging, and high-risk screening of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled and eligible to receive a contrast-enhanced breast MRI at the UMN Center for Clinical Imaging Research for either standard clinical care, or participation in the ISPY2/ACRIN6698 clinical research study
* Age 18 years or older
* Ability to read and understand English
* Ability to provide written informed consent

Exclusion Criteria:

* Subjects who are unlikely to tolerate the longer MRI scanning duration. This may include, history of discomfort during MRI scanning, anxiety, or claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients: recruited from the group of patients that have a known cancer and are scheduled to receive a breast MRI at the UMN Center for Clinical Imaging Research (CCIR)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Concentration of choline-containing metabolites | Baseline
  Demonstration of the feasibility of using SLIM-based techniques for acquiring spectoscopic data for quantifying choline and other metabolites in breast cancer.

SECONDARY OUTCOMES:
The apparent diffusion coefficient and T2 relaxation rate of water in the tumor | Baseline and 6 months following treatment
  Develop and optimize methods for performing diffusion weighted imaging and T2 relaxometry in breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Bolan, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Center for Clinical Imaging Reserach, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided